CLINICAL TRIAL: NCT05601271
Title: Effect of Allopurinol on Markers of Mineral and Bone Metabolism in Patients in With Chronic Kidney Disease: a Randomized Double-blind Study
Brief Title: Effect of Allopurinol on Markers of Mineral and Bone Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rosilene Motta Elias Coelho, MD, Ph.D, assistent nephrologist, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Alopurinol-CKD-MBD
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases; Osteodystrophy; Uric Acid Concentration, Serum, Quantitative Trait Locus 7
Keywords: chronic kidney disease; allopurinol; mineral and bone metabolism; uric acid; vitamin D
MeSH Terms: conditions — Renal Insufficiency, Chronic; Calcinosis | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): pills exactly as the drug will be delivered to participants. Instructions will be made to take the pill once a day.
  Interventions: Drug: Allopurinol
- Allopurinol (Active Comparator): pills exactly as the placebo will be delivered to participants. Instructions will be made to take the pill once a day.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol 100 to 300 mg a day for 3 months

SUMMARY:
Hyperuricemia is a common condition in patients with chronic kidney disease (CKD) in the glomerular filtration rate. Recently, it has been suggested that uric acid is related to a mineral and bone disease of CKD (CKD-MBD) since the high concentration of uric acid is associated with the harmful effect of vitamin D. The proof of concept of the association between acid uric acid and CKD-MBD is based on a prospective study (sample size 6) that observed, after 1 week of use of allopurinol, an increase in the concentration of 1,25(2D, a result independent of the concentration of calcium, phosphorus, 25(OH)D and PTH. An experimental study found that hyperuricemia could modify the expression of the 1α-hydroxylase enzyme, consequently reducing 1,25(OH). The current study aims to evaluate the action of allopurinol on CKD-MBD biomarkers (25(OH)-vitamin D, 1,25(OH)2D, FGF-23, PTH, calcium and phosphorus). We hypothesize that allopurinol can improve serum levels of 1,25(OH) 2D and PTH. This is a controlled, randomized, double-blind study, defined as a filtration rate < 60ml/1.73 m², according to the CKD-EPI equation. Inclusion criteria: patients with stages III, IV and V CKD who are not on dialysis with a serum level of 25(OH)-vitamin D >20 ng/ml. Exclusion criteria: Patients diagnosed with gout, undergoing treatment with allopurinol, patients already in use and drugs with sensitivity to the drug. Based on a previous study, we calculated a sample for 2 groups (placebo and drug) with pre and post-measurements (a total of 4). Considering a standard deviation of 4 and a difference of 7 in the treated group, 3 in the placebo group, and an alpha error of 5%, we calculated a sample of 25 patients in each arm.

DETAILED DESCRIPTION:
In this randomized double-blind study, patients receive allopurinol or a placebo for 3 months.

Dependent variables: 25(OH)-vitamin D, 1,25(OH)2D, FGF-23, PTH, calcium and phosphorus Population: stage 3, 4 or 5 CKD on conservative management at the Nephrology Service of Hospital das Clinicas HCFMUSP, Sao Paulo, Brazil.

The same physician will follow patients. Adverse effects will be recorded.

ELIGIBILITY:
Inclusion Criteria: stage 3, 4 or 5 CKD on conservative management

-

Exclusion Criteria:

* allergy to allopurinol
* current treatment with allopurinol
* Gout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
1,25 dihydroxivitamin D | 3 months
  Increase in 1,25 dihydroxivitamin D
FGF-23 | 3 months
  Reduction of FGF-23
Klotho | 3 months
  Increase in alpha Klotho

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided